CLINICAL TRIAL: NCT06798116
Title: Assessment of Liquid Platelet-Rich Fibrin Mixed With Denaturated Albumin Gel (ALB-PRF) or With Bone Allograft in The Treatment of Periodontal Intrabony Defects( Randomized Controlled Clinical Trial)
Brief Title: Treatment of Periodontal Intrabony Defects With Liquid Platelet-Rich Fibrin Mixed With Denaturated Albumin Gel (ALB_PRF)
Acronym: ALB-PRF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A04011023OM
Record Dates: First submitted 2024-11-05; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Bone Loss; Periodontitis Stage III; Intra-bony Pockets
Keywords: ALB-PRF; intrabony defect; periodontitis
MeSH Terms: conditions — Alveolar Bone Loss; Periodontitis | interventions — Fluid Therapy; Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: surgery and give medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- open flap debridement and demineralized freeze-dried bone allograft and mixed with liquid (PRF) (Experimental): will include 7 patients, in which the intrabony periodontal defects will be treated with open flap debridement and demineralized freeze-dried bone allograft (DFDBA) and mixed with liquid (PRF).
  Interventions: Procedure: Experimental: open flap debridement and demineralized freeze-dried bone allograft and mixed with liquid (PRF
- liquid (PRF) mixed with denatured albumin gel (ALB-PRF) injected in periodontal intrabony defects (Experimental): will include 7 patients, in which participants will be treated with open flap debridement and liquid (PRF) mixed with denatured albumin gel (ALB-PRF) will be injected in periodontal intrabony defects.
  Interventions: Procedure: defects will be treated with open flap debridement and liquid (PRF) mixed with denatured albumin gel (ALB-PRF) will be injected in periodontal intrabony defects
- open flap debridement, DFDBA mixed with liquid (PRF) and collagen membrane. (Active Comparator): will include 7 patients, in which participants will be treated with open flap debridement, DFDBA mixed with liquid (PRF) and collagen membrane.
  Interventions: Procedure: defects will be treated with open flap debridement , DFDBA mixed with liquid (PRF) and collagen membrane
- open flap debridement, DFDBA mixed with liquid (PRF) and ALB-PRF membrane. (Experimental): will include 7 patients in which participants will be treated with open flap debridement, DFDBA mixed with liquid (PRF) and ALB-PRF membrane.
  Interventions: Procedure: open flap debridement , DFDBA mixed with liquid (PRF) and ALB-PRF membrane.

INTERVENTIONS:
Procedure: Experimental: open flap debridement and demineralized freeze-dried bone allograft and mixed with liquid (PRF — Drawing 9 ml of blood into plastic test tubes without anticoagulants and other additives. This is followed by a centrifugation process according to the protocol for liquid PRF by using centrifuge under 2700rpm for 8 min.
  The yellow top layer, formed upon centrifugation, consists of platelet-poor plasma that will be collect by a syringe in a volume of 2 ml, liquid PRF and buffy coat that will also be collected by a syringe in a volume of 4 ml. The Platelet-Poor plasma in the syringe will be transferred to a special machine that increases its temperature to 75°C for 10 minutes. ALB-PRF will be prepared by mixing the albumin gel with liquid concentrated growth factor including the buffy coat in a separate syringe by utilizing a female luer lock connector to obtain the injectable ALB-PRF in final ready form. in this group;, the defects will be treated with open flap debridement and DFDBA and mixed with liquid (PRF)
  Arms: open flap debridement and demineralized freeze-dried bone allograft and mixed with liquid (PRF)
Procedure: defects will be treated with open flap debridement and liquid (PRF) mixed with denatured albumin gel (ALB-PRF) will be injected in periodontal intrabony defects — Drawing 9 ml of blood into plastic test tubes without anticoagulants and other additives. This is followed by a centrifugation process according to the protocol for liquid PRF by using centrifuge under 2700rpm for 8 min.
  The yellow top layer, formed upon centrifugation, consists of platelet-poor plasma that will be collect by a syringe in a volume of 2 ml, liquid PRF and buffy coat that will also be collected by a syringe in a volume of 4 ml. The Platelet-Poor plasma in the syringe will be transferred to a special machine that increases its temperature to 75°C for 10 minutes. ALB-PRF will be prepared by mixing the albumin gel with liquid concentrated growth factor including the buffy coat in a separate syringe by utilizing a female luer lock connector to obtain the injectable ALB-PRF in final ready form. in this group;, defects will be treated with open flap debridement and liquid (PRF) mixed with denatured albumin gel (ALB-PRF) will be injected in periodontal intrabony defects.
  Arms: liquid (PRF) mixed with denatured albumin gel (ALB-PRF) injected in periodontal intrabony defects
Procedure: defects will be treated with open flap debridement , DFDBA mixed with liquid (PRF) and collagen membrane — Drawing 9 ml of blood into plastic test tubes without anticoagulants and other additives. This is followed by a centrifugation process according to the protocol for liquid PRF by using centrifuge under 2700rpm for 8 min.
  The yellow top layer, formed upon centrifugation, consists of platelet-poor plasma that will be collect by a syringe in a volume of 2 ml, liquid PRF and buffy coat that will also be collected by a syringe in a volume of 4 ml. The Platelet-Poor plasma in the syringe will be transferred to a special machine that increases its temperature to 75°C for 10 minutes. ALB-PRF will be prepared by mixing the albumin gel with liquid concentrated growth factor including the buffy coat in a separate syringe by utilizing a female luer lock connector to obtain the injectable ALB-PRF in final ready form. in this group;, the defects will be treated with open flap debridement , DFDBA mixed with liquid (PRF) and collagen membrane
  Arms: open flap debridement, DFDBA mixed with liquid (PRF) and collagen membrane.
Procedure: open flap debridement , DFDBA mixed with liquid (PRF) and ALB-PRF membrane. — Drawing 9 ml of blood into plastic test tubes without anticoagulants and other additives. This is followed by a centrifugation process according to the protocol for liquid PRF by using centrifuge under 2700rpm for 8 min.
  The yellow top layer, formed upon centrifugation, consists of platelet-poor plasma that will be collect by a syringe in a volume of 2 ml, liquid PRF and buffy coat that will also be collected by a syringe in a volume of 4 ml. The Platelet-Poor plasma in the syringe will be transferred to a special machine that increases its temperature to 75°C for 10 minutes. ALB-PRF will be prepared by mixing the albumin gel with liquid concentrated growth factor including the buffy coat in a separate syringe by utilizing a female luer lock connector to obtain the injectable ALB-PRF in final ready form. in this group;, the defects will be treated with open flap debridement , DFDBA mixed with liquid (PRF) and ALB-PRF membrane.
  Arms: open flap debridement, DFDBA mixed with liquid (PRF) and ALB-PRF membrane.

SUMMARY:
The objective of study also is to assess radiographic linear defect depth, and radiographic defect bone density following the application of liquid Platelet-Rich Fibrin (PRF) mixed with denaturated Albumin gel (ALB-PRF) or with bone allograft in periodontal intrabony defects.

Patients and methods: 28 patients will be selected from the outpatient clinic in the Oral Medicine and Periodontology Department, Faculty of Dentistry, Mansoura University according to Pre-operative CBCT that will be used to evaluate the bone destruction pattern. According to the techniques that used in the treatment of periodontal bony defect, the participants will be randomly divided into 4 equal groups: Group I: will include 7 patients, in which the intrabony periodontal defects will be treated with open flap debridement and demineralized freeze-dried bone allograft (DFDBA) and mixed with liquid (PRF). Group II: will include 7 patients, in which participants will be treated with open flap debridement and liquid (PRF) mixed with denatured albumin gel (ALB-PRF) will be injected in periodontal intrabony defects. Group III: will include 7 patients, in which participants will be treated with open flap debridement, DFDBA mixed with liquid (PRF) and collagen membrane. Group IV: will include 7 patients in which participants will be treated with open flap debridement, DFDBA mixed with liquid (PRF) and ALB-PRF membrane.

DETAILED DESCRIPTION:
28 patients will be selected from the outpatient clinic in the Oral Medicine and Periodontology Department, Faculty of Dentistry, Mansoura University according to Pre-operative CBCT that will be used to evaluate the bone destruction pattern.

Sample size will be calculated using G-Power 3.1 for Mac with (α = 0.05, and power = 0.95). One-way ANOVA test will be used and effect size of (0.7) based on the anticipated mean difference of the efficacy of new generation platelet-rich fibrin according Nagy et.al 2021. The total sample size of the four groups will be 28 patients.

Inclusion criteria:

* periodontits stage III according to classification of periodontal and peri-implant disease and conditions (2018).
* Patient with two or three walls or combined bony defect.
* Favorable pattern of occlusion.
* Patient ability to comply with the required recall visits.

Exclusion Criteria:

* Local or systemic diseases that contraindicate surgery.
* Smokers
* Patients with parafunctional habits.
* Pregnancy or lactation.
* Diabetic patient.
* Osteoporosis.
* Immune-suppressed condition that may affect the outcome of the therapy.

I) Study design:

According to the techniques that used in the treatment of periodontal bony defect, the participants will be randomly divided into 4 equal groups:

Group I: will include 7 patients, in which the intrabony periodontal defects will be treated with open flap debridement and demineralized freeze-dried bone allograft (DFDBA) and mixed with liquid (PRF).

Group II: will include 7 patients, in which participants will be treated with open flap debridement and liquid (PRF) mixed with denatured albumin gel (ALB-PRF) will be injected in periodontal intrabony defects.

Group III: will include 7 patients, in which participants will be treated with open flap debridement, DFDBA mixed with liquid (PRF) and collagen membrane.

Group IV: will include 7 patients in which participants will be treated with open flap debridement, DFDBA mixed with liquid (PRF) and ALB-PRF membrane.

II) Surgical Procedures ,liquid PRF and ALB-PRF preparation:

Patients will be premedicated by Amoxicillin 2 gm one hour before surgery as a prophylactic antibiotic, in addition patient will instructed to rinse with a 0.2% chlorhexidine mouth wash for 1 minute immediately prior to surgery.

All patients will be subjected to surgical procedure consisting of the injection of local anaesthetic Articaine hydrochloride 4% with epinephrine (1:100,000) followed by sulcular incision with 15c blade, reflection of a full thickness flap atraumaticlly , open flap debridement using periodontal curettes to remove all tissue tags and granulation tissue. Ethylenediaminetetraacetic acid (EDTA) will be applied to the root surface followed by rinsing with normal saline.

Liquid (PRF) and ALB-PRF Preparation:

As the protocol entails drawing 9 ml of blood into plastic test tubes without anticoagulants and other additives. This is followed by a centrifugation process according to the protocol for liquid PRF by using centrifuge under 2700rpm for 8 min.

The yellow top layer, formed upon centrifugation, consists of platelet-poor plasma that will be collect by a syringe in a volume of 2 ml, liquid PRF and buffy coat that will also be collected by a syringe in a volume of 4 ml. The Platelet-Poor plasma in the syringe will be transferred to a special machine that increases its temperature to 75°C for 10 minutes. ALB-PRF will be prepared by mixing the albumin gel with liquid concentrated growth factor including the buffy coat in a separate syringe by utilizing a female luer lock connector to obtain the injectable ALB-PRF in final ready form.

In group I, the defects will be treated with open flap debridement and DFDBA and mixed with liquid (PRF). In group II, the defects will be treated with open flap debridement and liquid (PRF) mixed with denatured albumin gel (ALB-PRF) will be injected in periodontal intrabony defects. In group III, the defects will be treated with open flap debridement , DFDBA mixed with liquid (PRF) and collagen membrane. In group IV, the defects will be treated with open flap debridement, DFDBA mixed with liquid (PRF) and ALB-PRF membrane. Vertical mattress suture with 5-0 suture will be used to close the wound.

Patients will be instructed to use 0.2% chlorhexidine gluconate mouth wash for 1 minute twice a day for 2 weeks, also maintained on amoxicillin 1gm twice a day for six days postoperatively and Ibuprofen 400 mg will be prescribed to be taken 2 to 4 times a day during meals as analgesic.

Clinical assessment: Pain and bruising will be obtain using Visual Analogue Scales (VAS) on days 0, 3, 5 and 7 post-operatively. While healing will be assess at days 2,7 and 14. The following periodontal indices will be assessed at baseline, 3 and 6 months: Plaque index (PI). Bleeding on Probing (BOP). Pocket depth (PD). Clinical Attachment Level (CAL). Radiographic Assessment: Using cone beam CT (CBCT) scan to assess linear bone defect depth and defect bone density at baseline and 6 months.

Statistical analysis: The data will be collected and statistical analysis will be done using SPSS(statistical package for social sciences) version 2024.

ELIGIBILITY:
Inclusion Criteria:

* Periodontist stage III according to classification of periodontal and peri-implant disease and conditions (2018).
* Patient with two or three walls or combined bony defect.
* Favourable pattern of occlusion.
* Patient ability to comply with the required recall visits.

Exclusion Criteria:

* Local or systemic diseases that contraindicate surgery.
* Smokers
* Patients with parafunctional habits.
* Pregnancy or lactation.
* Diabetic patient.
* Osteoporosis.
* Immune-suppressed condition that may affect the outcome of the therapy.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-01-24 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
pocket depth | pocket depth will be assessed at baseline, 3 and 6 months.
  pocket depth: by placing dental probe between your teeth and gumline. Pockets are measured at several places in your upper and lower gums. In a healthy mouth, the pocket depth is usually between 1 and 3 millimetres (mm). Pockets deeper than 4 mm may indicate periodontitis
Plaque index | At baseline ,3and 6 months
  Evaluation of existence plaque in all around tooth aspects
Bleeding on Probing | At baseline ,3 and 6months.
  Evaluation of existence Bleeding during gentle periodontal probing.
Clinical Attachment Level | At baseline ,3 and 6 months.
  To assess the clinical attachment level.

SECONDARY OUTCOMES:
Pain score | At day 0,3,5 and 7 post-operatively. While healing will be assess at days 2,7 and 14
  The patients will report their pain score directly through VAS score (between 0 and 10; 0: no pain, 1: minimal pain, 5: moderate pain, and 10: severe pain).
Alveolar ridge width (buccolingual). | At base line and 6 months starting from base line.
  Will be assessed via Cone-Beam Computed Tomography (CBCT) that Provides a radiographic assessment of the buccolingual width by measuring the distance between buccal and lingual bone walls.
Alveolar ridge height (apicocronal) | At base line and 6 months starting from base line.
  Will be assessed via Cone-Beam Computed Tomography (CBCT) that Provides a radiographic assessment of the apicocronal height by measuring the ridge height from the top of the alveolar ridge to the upper border of the alveolar canal.
Bone density | At base line and 6 months starting from base line.
  Will be assessed via Cone-Beam Computed Tomography (CBCT) The measurement helps in assessing the quality of bone directly through Hounsfield units (HU) (between D1 and D5; D1: > 1250 HU, D2: 850 to 1250 HU, D3: 350 to 850 HU, D4: 150 to 350 HU, D5: < 150 HU).

CONTACTS AND LOCATIONS:
Overall Officials: Dhaidan Naif Alshammari, Bachelor, Principal Investigator — faculty of dentistry Mansoura university
Locations (1):
- faculty of dentistry Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
after Completing the study ; the data will be available when requested